CLINICAL TRIAL: NCT00653796
Title: SCH 58235: A Multicentre, Randomised, Parallel Group, Placebo-Controlled Study Comparing the Efficacy, Safety, And Tolerability of the Daily Co-Administration of Ezetimibe 10 mg With Atorvastatin 10 mg vs. Ezetimibe Placebo With Atorvastatin 10 mg in Untreated Subjects With Primary Hypercholesterolaemia and Coronary Heart Disease
Brief Title: Ezetimibe Plus Atorvastatin Versus Atorvastatin in Untreated Subjects With High Cholesterol (P03434)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Organon and Co (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P03434
Record Dates: First submitted 2008-04-01; First posted 2008-04-07 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Hypercholesterolemia; Atherosclerosis
MeSH Terms: conditions — Hypercholesterolemia; Atherosclerosis | interventions — Ezetimibe; Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ezetimibe + Atorvastatin (Experimental)
  Interventions: Drug: Ezetimibe + Atorvastatin
- Atorvastatin (Active Comparator)
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Ezetimibe + Atorvastatin — oral tablets: ezetimibe 10 mg + atorvastatin 10 mg once daily for 6 weeks
  Other Names: SCH 58235; Zetia; Lipitor
  Arms: Ezetimibe + Atorvastatin
Drug: Atorvastatin — oral tablets: atorvastatin 10 mg + ezetimibe placebo once daily for 6 weeks
  Other Names: Lipitor
  Arms: Atorvastatin

SUMMARY:
This study was designed to assess whether co-administration of ezetimibe 10 mg with atorvastatin 10 mg in treatment naïve subjects would be more effective than treatment with atorvastatin 10 mg alone for reducing LDL-concentrations.

ELIGIBILITY:
Inclusion Criteria:

* Male and non-pregnant female subjects, who demonstrated willingness to participate and comply with procedures by signing informed consent, and who were >=18 years and <=75 years of age, were eligible to participate if they had: a baseline LDL-C concentration >=3.3 mmol/L (130 mg/dL) to <=4.9 mmol/L (190 mg/dL); a baseline triglyceride concentration of <3.99 mmol/L (350 mg/dL); a documented history of coronary heart disease (CHD); a stable weight history for 4 weeks prior to baseline; completion of the designated washout periods for all prohibited medications; and did not fulfill any of the exclusion criteria for the study.

Exclusion Criteria:

* Body Mass Index of >=30 kg/m^2 at baseline (increased to 35 kg/m^2 in protocol amendment 1
* Liver transaminase (ALT, AST) >1.5 times the upper limit of normal and with no active liver disease at baseline
* Evidence of current myopathy (excluding subjects with CK >1.5 times above the upper limit of normal at baseline
* Clinical lab tests (CBC, blood chemistries, urinalysis) results outside the normal range or unacceptable to the investigator at baseline
* Type II diabetes mellitus that was poorly controlled (HbA1c>9%), newly diagnosed, or changed their anti-diabetic therapy within 3 months of baseline
* Type I diabetes mellitus and not on a stable insulin regimen for 3 months prior to baseline or who had a recent history of repeated hypoglycaemia or unstable glycaemic control
* Known hypersensitivity to HMG-CoA reductase inhibitors
* Alcohol consumption >14 units (women)/21 units (men) (unit = 0.5 pint of beer or wine, or single measure of spirits)
* Pregnancy, lactation, or any condition or situation which, in the opinion of the investigator, posed a risk to the subject or interfered with participation in this study.
* Any of the following medical conditions: HIV positive; congestive heart failure defined by NYHA as Class III or IV; uncontrolled cardiac arrhythmia; MI, acute coronary insufficiency, CABG, or angioplasty within 3 months of baseline; unstable or severe peripheral artery disease within 3 months of baseline; newly diagnosed or unstable angina pectoris at baseline; uncontrolled hypertension with systolic blood pressure >100 mm Hg at baseline; uncontrolled endocrine or metabolic disease known to influence serum lipids or lipoproteins; impaired renal function or nephritic syndrome at baseline; disorders of the hematological, gastrointestinal, or central nervous systems; diseases other than hyperlipidaemia or coronary heart disease that would have interfered with study evaluations; and cancer.
* Drug abuse or emotional or intellectual problems;
* Use of certain drugs, food, or other agents known to alter cholesterol levels or to cause pharmacokinetic interactions with either ezetimibe or atorvastatin

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2003-09-01 (Actual); Primary Completion 2004-08-01 (Actual); Study Completion 2004-08-01 (Actual)

PRIMARY OUTCOMES:
Percent change in LDL-C from baseline to endpoint. | 6 weeks

SECONDARY OUTCOMES:
Percent change from baseline to endpoint in total cholesterol, HDL-C and triglycerides. | 6 weeks
Safety: adverse events, laboratory test results, vital signs. | Throughout study

REFERENCES:
- [Result] Blagden MD, Chipperfield R. Efficacy and safety of ezetimibe co-administered with atorvastatin in untreated patients with primary hypercholesterolaemia and coronary heart disease. Curr Med Res Opin. 2007 Apr;23(4):767-75. doi: 10.1185/030079907x182059. PMID 17407633